CLINICAL TRIAL: NCT06909591
Title: Transcultural and Psychometric Validation of the Lubben Social Network Scale in Older Adults Living in the French West Indies
Acronym: VALLUB
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital Center of Martinique (Other)
Responsible Party: Sponsor
Other Study IDs: 24_RIPH3-05; 2024-A02609-38 (Registry Identifier: ID-RCB)
Record Dates: First submitted 2025-03-27; First posted 2025-04-03 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-03

CONDITIONS: Geriatric Assessment; Patients Over 65 Years Old
Keywords: Geriatrics; Lubben Social Network Scale; Transcultural validation; Psychometric validation; Martinique; French West Indies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients aged 65 or older: For the transcultural validation, a french version of the Lubben Social Network Scale questionnaire will be produced. For the psychometric validation, 150 patients aged of 65 or older will pass the questionnaire. The Duke Health Profile questionnaire will be also passed by the subject, for the convergent validity.
  Interventions: Other: Self-assessment questionnaire

INTERVENTIONS:
Other: Self-assessment questionnaire — 150 patients aged of 65 or older will pass the Lubben Social Network Scale questionnaire. The Duke Health Profile questionnaire will be also passed by the subject, for the convergent validity.

SUMMARY:
Social isolation and loneliness are common among older adults. They are associated with high morbidity and mortality, with an impact comparable to that of other known risk factors such as obesity, a sedentary lifestyle, smoking, etc.

To date, there is no tool to measure social isolation and loneliness for patients living in the French West Indies. Applying unadapted and unvalidated tools to them without taking into account local ethnocultural realities would be risky.

The investigators believe it is necessary to adapt the scales used to measure social isolation and loneliness for a population living in the French West Indies.

Through this study, the investigators propose adapting the Lubben Social Network Scale, a social isolation questionnaire, for this population and conducting its psychometric validation.

DETAILED DESCRIPTION:
Social isolation and loneliness are common among older adults. They are associated with high morbidity and mortality, with an impact comparable to that of other known risk factors such as obesity, a sedentary lifestyle, smoking, etc.

Loneliness is a subjective concept of social relationships, most often reflecting a negative feeling.

Social isolation, on the other hand, is an objective concept of social relationships and refers to infrequent or rare contact with family and friends and can also include living alone.

The feeling of loneliness is linked to social isolation, although the association is only partial.

Indeed, some socially isolated people do not always experience loneliness; and some people living alone are not always socially isolated.

Two theories of loneliness argue that a mismatch between expectations and realities of social contact (cognitive theory) and a lack of intimate or social relationships (deficit theory) can lead to feelings of social or emotional loneliness.

A meta-analysis showed that the risk of premature death was 26% higher in people experiencing loneliness, 29% higher in those who were socially isolated, and 32% higher in the group living alone.

Another meta-analysis examined the effects of loneliness and social isolation on (among other things) mortality. The results showed that loneliness and social isolation were significantly associated with an increased risk of mortality.

The authors conclude that further research is needed to confirm whether loneliness and social isolation have a direct impact on mortality, or whether the association is indirect via the cardiovascular system and psychological health.

To date, there is no tool to measure social isolation and loneliness for patients living in the French West Indies. Applying unsuitable and unvalidated tools to them without taking into account local ethnocultural realities would be risky.

The investigators believe it is necessary to adapt the scales used to measure social isolation and loneliness for a population living in the French West Indies.

Through this study, the investigators propose adapting the Lubben Social Network Scale, a social isolation questionnaire, for this population and conducting its psychometric validation.

ELIGIBILITY:
Inclusion Criteria:

* Patient ≥ 65 years old,
* Hospitalized (Geriatric Day Hospital (HDJ) or Geriatric Medical Care and Rehabilitation Service (SMT)), or seen in geriatric external consultation,
* MMS ≥ 20,
* Patient able to understand and answer a self-administered questionnaire in French,
* Patient having been informed of the research,
* Patient agreeing to participate in the study.

Exclusion Criteria:

* Patient with sensory disorders preventing completion of the questionnaire,
* Patient unable to consent to participate in the study,
* Patient under legal protection, guardianship, or curatorship,
* Patient who has refused to participate in the study.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients aged of 65 or older
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Transcultural validation of the Lubben Social Network Scale questionnaire | 1 month
  It will be a question of obtaining a version translated into French. The translated version tested on a small group of patients (15-40) will be submitted to the author of the original version of the tool, along with a report highlighting and explaining all the modifications and difficulties noted by a group of experts.
Psychometric validation of the Lubben Social Network Scale questionnaire | 24 months
  Questionnaire will be passed by 150 subjects. Following parameters will be measured: feasibility and acceptability, validity, reliability, and sensitivity to change.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU of Martinique, Fort-de-France, Martinique

IPD SHARING:
Plan to Share IPD: No